CLINICAL TRIAL: NCT01800994
Title: Multicenter, Prospective, Observational, Non Interventional Clinical Trial to Assess the Asthma and COPD Treatment by Inhalation Devices
Brief Title: Prospective evAluatIon foR Inhalation Devices Study
Acronym: PAIR
Status: Completed | Type: Observational
Sponsor: Elpen Pharmaceutical Co. Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2012-HAL-EL-32
Record Dates: First submitted 2013-02-20; First posted 2013-02-28 (Estimated); Last update posted 2021-04-12 (Actual); Status verified 2014-08

CONDITIONS: Asthma; COPD
Keywords: convenience
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- asthma, COPD: patients with asthma and COPD treated with inhalation devices

SUMMARY:
ASTHMA:

Asthma is a chronic inflammatory disorder of the airways in which many different types of cells, and various cellular components. The chronic inflammation causes an increase of the over-responsiveness of the airways, which leads to recurrent episodes of wheezing, breathlessness, chest tightness, and coughing, particularly at night or in the early morning hours. These episodes, usually associated with widespread but variable block the airway, which is usually reversible either spontaneously or by treatment.

Asthma is one of the most common chronic diseases worldwide, posing significant social burden in both children and adults. It is estimated that about 300 million people currently suffer from asthma. The incidence of asthma is universal regardless of the level of development of the country. There is evidence that over the last 20 years the prevalence has increased significantly, specially in pediatric populations.

COPD:

Chronic Obstructive Pulmonary Disease (COPD) is a major public health problem. It is the fourth leading cause of chronic morbidity and mortality in the United States after heart disease, strokes and acute respiratory infections, while on an annual basis, the disease robs the lives of more than 3,000,000 people around us worldwide. The most worrying is that the impact has been steadily rising, and this dramatic increase in the frequency shows that by 2020 the disease will be the third leading cause of death. In Greece, 8.4% of the population suffers from COPD.

Smoking is the leading cause of COPD. However, not all smokers develop the clinical picture of COPD, suggesting that additional factors are involved in manifestation. Further investigation of risk factors for COPD, methods of reducing exposure to these agents and the molecular and cellular mechanisms involved in the pathogenesis remain a major area of research to develop effective treatments that will reduce or prevent the development the disease.

DETAILED DESCRIPTION:
ASTHMA TREATMENT:

As regards the pharmacological management of asthma, inhaled corticosteroids (eg budesonide, fluticasone and beclomethasone) underlying the maintenance therapy, while beta-2 agonists are the long-term preferred additional treatment. Other common medications are systemic corticosteroids, beta-2-agonist short duration (eg salbutamol) oral beta2-agonists, long-lasting, methylxanthines, converters leukotrienes, colors and anticholinergics.

The main clinical advantages of transport and deposition of the drug directly to the lungs associated with the safety and efficacy: the side effects associated with the systemic circulation zero, while high concentrations of the active substance can be directly attributed to the points of action. Furthermore, the onset of action of inhaled beta2-agonist is faster that of oral beta-2 agonist and the therapeutic response is achieved faster. Finally, require lower doses of the drug, due to the efficiency of this direct lungs, reducing the problems of poor absorption and metabolism by the liver.

COPD TREATMENT:

Effective management of COPD involves four steps: (1) assessment and monitoring of the disease, (2) minimize the risk factors, (3) stabilization of disease, and (4) the treatment of an exacerbation.

ELPENHALER:

A new multi-single dose inhaled dry powder (Elpenhaler ®) has been designed, developed and patented by the Elpen Pharmaceutical Co. Inc (Pikermi, Greece). The new inhaler is suitable for the performance of a range of drugs for asthma, such as budesonide, formoterol and fluticasone.

OTHER TREATMENT APPROACHES:

Most asthma medications are administered in the form of inhalers. There are various forms of devices that facilitate the administration of inhaled medications in young children. The correct use of inhalers drugs is very important for the treatment of asthma. If the patient does not understand the correct instructions, the drug is deposited satisfactorily lungs, ie organ must act, so there is no remission. Furthermore when the inhalers incorrectly used much of the drug remains in the oral cavity and the pharynx and therefore the patient is exposed to any adverse events drug while not treated properly asthma. Appropriate for patient inhaler should be chosen by the attending physician, after confirmation by pilot demonstration site at the clinic, the patient (depending on age) have understood and can apply the device user. A new study conducted by the Center for Capital allergies and respiratory diseases showed that 25% of asthmatic subjects reported that the inhaler was empty during an asthma attack. The reason: "There is no way for someone to see how much medicine has used the inhaler continues to blow air even when it is empty," says Bradley Chips, who was lead author of the study. To save your breath, look at the package leaflet number of inhaled doses contain.

ELIGIBILITY:
Inclusion Criteria:

* Patients (newly diagnosed or not) with asthma and / or COPD, who use correctly (according to the opinion of the responsible investigator) their device
* Male or female patients aged 18 years
* Patients with compliance to treatment
* Patients with compliance to the study procedures
* Patients who have signed the study participation consent form.

Exclusion Criteria:

* Patients who use incorrectly their inhalational devices
* Male or female patients under 18 years
* Patients who are non-compliant to their treatment for asthma and COPD
* Patients who are non-compliant to study procedures
* Patients who have not signed the study participation consent form.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Asthma and COPD treated by inhalation devices
Sampling Method: Non-Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2013-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
FSI-10 score | 2 months treatment
  FSI-10 questionnaire total score FSI-10 questionnaire score per question

SECONDARY OUTCOMES:
Adverse Events Reporting | 2 months treatment
  Number of Adverse Events occured during study duration.

CONTACTS AND LOCATIONS:
Overall Officials: Spyridon Papiris, MD, Professor, Study Director — Professor of Pulmonology, Attikon University Hospital of Athens; Athina Vlachou, MD, Principal Investigator — Private Office; Areti Xifteri-Nikolinati, MD, Principal Investigator — Messini, Greece; Georgios Efraimidis, MD, Principal Investigator — Plmonology Hospital of Patras, Greece; Nikolaos Harokopos, MD, Principal Investigator — General hospital of Pyrgos, Peloponnese, Greece; Dionysia Kalampoka, MD, Principal Investigator — Private Office, Patras, Greece; Athanasia Christara, MD, Principal Investigator — Private Office, Korinthos, Greece; Emmanouel Fothiantakis, MD, Principal Investigator — Private Office, Chaidari, Athens, Greece; Elias Kainis, MD, Principal Investigator — Sotiria Pulmonogy Hospital of Athens; Adamantia Liapikou, MD, Principal Investigator — Sotiria Pulmonary Hospital of Athens; Xenophon Agelidis, MD, Principal Investigator — Attikon Hospital; Antonios Kopanakis, MD, Principal Investigator — Thriasio General Hospital, Greece; Konstantina Houliara, MD, Principal Investigator — Private office, Patisia, Athens, Greece; Helen Adamou, MD, Principal Investigator — Nea Filadelfia, Athens, Greece; George Kalfountzos, MD, Principal Investigator — Private office, Larissa, Greece; Athanasios Pitenis, MD, Principal Investigator — Private Office, Grevena, Greece; Eugeneia Karyanou, MD, Principal Investigator — Private Office, Kaisariani, Athens, Greece; Georgia Kotantoula, MD, Principal Investigator — Private Office, Gerakas, Attika, Greece; Evangelos Bourantzis, MD, Principal Investigator — Private office, Athens, Greece; Konstantinos Marosis, MD, Principal Investigator — Sotiria Pulmonary Hospital of Athens; Harilaos Lambrakis, MD, Principal Investigator — Sotiria Pulmonary Hospital of Athens; Anastasios Palamidas, MD, Principal Investigator — Sotiria Pulmonary Hospital of Athens; Dimitrios Zois, MD, Principal Investigator — General Hospital of Karditsa, Greece; Maria Varouha, MD, Principal Investigator — Private office, Rethymno, Crete, Greece; Karmen Stahouli, MD, Principal Investigator — Hatzikosta Hospital of Ioannina, Greece; Peter Oikonomides, MD, Principal Investigator — General Hospital of Filiata, Thesprotia, Greece; George Balasoulis, MD, Principal Investigator — Private office, Thessaloniki, Greece; Konstantinos Porpodis, MD, Principal Investigator — Private office, Thessaloniki, Greece; Despina Melemeni, MD, Principal Investigator — Sismanogleio Hospital of Athens, Greece; Andreas Stratis, MD, Principal Investigator — Private office, Greece; Efrosini Manali, MD, Principal Investigator — Attikon University Hospital of Athens, Greece; Theodora Tsiounta, MD, Principal Investigator — Theageneio oncology hospital of Thessaloniki, Greece; Anna Gavriilidou, MD, Principal Investigator — Papageorgiou hospital of Thessaloniki, Greece; Athanasia Pataka, MD, Principal Investigator — Papanikolaou General hospital of Thessaloniki, Greece; Chrysavgi Terovitou, MD, Principal Investigator — General hospital of Kavala, Greece; Elisavet Christina Filippidou, MD, Principal Investigator — General hospital of Kavala, Greece; Paschalis Kakavelas, MD, Principal Investigator — Private office, Piraeus, Greece; Nikolaos Manolakoglou, MD, Principal Investigator — Private office, Kalamaria, Thessaloniki, Greece; Evangelia Tsikrika, MD, Principal Investigator — General hospital of Veroia, Greece; Athanasios Papandreou, MD, Principal Investigator — Private office, Orestiada, Greece; Vasilios Adamidis, MD, Principal Investigator — Private office, Kozani, Greece; Paraskevi Tsafaridou, MD, Principal Investigator — Private office, Thessaloniki, Greece; Maria Katertzi, MD, Principal Investigator — Private office, Moudania, Thessaloniki, Greece; Pashalia Tsiaga, MD, Principal Investigator — Private office, Serres, Greece; Christos Babalis, MD, Principal Investigator — Private office, Serres, Greece; Konstantinos Albantakis, MD, Principal Investigator — Private office, Larisa, Greece; Martha Andritsou, MD, Principal Investigator — Sotiria Pulmonology Hospital of Athens
Locations (6):
- Greece (6):
  - Evagelismos hospital, Athens
  - Private Office, Athens
  - General State hospital of Lamia, Lamia
  - Private Office, Piraeus
  - Private Office, Volos
  - Asklipiion Hospital, Voula

REFERENCES:
- [Background] Reliability of the FSI-10 questionnaire for the assessment of the usability of drug inhalers in Greek patients, accepted for publication by 'Archives of Hellenic Medicine'
- [Background] Global Strategy for Asthma Management and Prevention NIH Publication No 02-3659 Issued January, 1995 (updated 2002) Management Segment (Chapter 7): Updated 2005 from the 2004 document. The GINA reports are available on www.ginasthma.org
- [Background] British Thoracic Society; Scottish Intercollegiate Guidelines Network. British guideline on the management of asthma. Thorax. 2003 Feb;58 Suppl 1(Suppl 1):i1-94. doi: 10.1136/thorax.58.suppl_1.1i. No abstract available. PMID 12653493
- [Background] National Asthma Education and Prevention Program. National Asthma Education and Prevention Program. Expert Panel Report: Guidelines for the Diagnosis and Management of Asthma Update on Selected Topics--2002. J Allergy Clin Immunol. 2002 Nov;110(5 Suppl):S141-219. No abstract available. PMID 12542074
- [Background] National Institutes of Health. Global strategy for asthma management and prevention. Bethesda (MD): Global Initiative for Asthma (GINA), National Institutes of Health, 2002 Feb. Publication no. 02-3659
- [Background] Dolovich MA, MacIntyre NR, Anderson PJ, Camargo CA Jr, Chew N, Cole CH, Dhand R, Fink JB, Gross NJ, Hess DR, Hickey AJ, Kim CS, Martonen TB, Pierson DJ, Rubin BK, Smaldone GC. Consensus statement: aerosols and delivery devices. American Association for Respiratory Care. Respir Care. 2000 Jun;45(6):589-96. No abstract available. PMID 10894452
- [Background] ICH topic E9 statistical principles for clinical trials - Note for guidance on statistical principles for clinical trials (CPMP/ICH/363/96).
- [Background] Frey U, Stocks J, Coates A, Sly P, Bates J. Specifications for equipment used for infant pulmonary function testing. ERS/ATS Task Force on Standards for Infant Respiratory Function Testing. European Respiratory Society/ American Thoracic Society. Eur Respir J. 2000 Oct;16(4):731-40. doi: 10.1034/j.1399-3003.2000.16d28.x. PMID 11106221
- [Background] van Beerendonk I, Mesters I, Mudde AN, Tan TD. Assessment of the inhalation technique in outpatients with asthma or chronic obstructive pulmonary disease using a metered-dose inhaler or dry powder device. J Asthma. 1998;35(3):273-9. doi: 10.3109/02770909809068218. PMID 9661680
- [Background] Campbell JL, Kiebert GM, Partridge MR. Development of the satisfaction with inhaled asthma treatment questionnaire. Eur Respir J. 2003 Jul;22(1):127-34. doi: 10.1183/09031936.03.00097503. PMID 12882462
- [Background] Lenney J, Innes JA, Crompton GK. Inappropriate inhaler use: assessment of use and patient preference of seven inhalation devices. EDICI. Respir Med. 2000 May;94(5):496-500. doi: 10.1053/rmed.1999.0767. PMID 10868714
- [Background] van der Palen J, Klein JJ, van Herwaarden CL, Zielhuis GA, Seydel ER. Multiple inhalers confuse asthma patients. Eur Respir J. 1999 Nov;14(5):1034-7. doi: 10.1183/09031936.99.14510349. PMID 10596686
- [Background] Perpina Tordera M, Viejo JL, Sanchis J, Badia X, Cobos N, Picado C, Sobradillo V, Martinez Gonzalez del Rio J, Duce F, Munoz Cabrera L. [Assessment of patient satisfaction and preferences with inhalers in asthma with the FSI-10 Questionnaire]. Arch Bronconeumol. 2008 Jul;44(7):346-52. Spanish. PMID 18727886
- [Background] Global Initiative for Chronic Obstructive Lung Disease, Global Strategy for the Diagnosis, Management and Prevention of Cronic Obstructive Pulmonary Disease (Updated 2009)